CLINICAL TRIAL: NCT01662596
Title: Detection of Risk Factors for Fetal Anomalies in a Rural Hospital Population
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0044-12-HYMC
Record Dates: First submitted 2012-08-07; First posted 2012-08-10 (Estimated); Last update posted 2012-08-10 (Estimated); Status verified 2012-08

CONDITIONS: Pregnancy; Pregnancy Complications
Keywords: Risk factors,; prenatal diagnosis,; fetal malformations
MeSH Terms: conditions — Pregnancy Complications; Congenital Abnormalities

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of the study is to estimate the rate of risk factors for appearance of disease or fetal malformations in a population who turn to hospital "Hillel Yaffe" and examine whether there is a difference in the rate of early testing for diseases or birth defects in the fetus.

Understanding the population and its risk factors, will allow specific reference to these risk factors to lowering them to eventually reduce the rate of congenital malformations in this population.

DETAILED DESCRIPTION:
Major defects prevalence in the general population is estimated at 5% of all live births. In cases where the fetus suffers from structural defect, chromosomal or genetic disease, prenatal diagnosis is an important scientific tool that allows reliable advice and better pregnancy outcomes.

Diseases and many embryonic defects can be detected early, including nervous system defects, heart defects, urinary tract defects, limb defects and more. Taking folic acid before pregnancy and during the first trimester reduces the incidence of some of these defects.

Aneuploidy and mainly trisomy 21,18,13, Monosomy X and aneuploid in sex chromosome is responsible for most of the chromosomal anomalies. Some of aneuploidy can be diagnosed by a combination of nuchal translucency (also associated with cardiac abnormalities) and maternal serum markers detection in the first trimester of pregnancy or a laboratory test in the second trimester. Ultrasound is also a tool for diagnosis of aneuploidity, which detecting abnormalities characteristic or "soft signs" who suspicious in chromosomal disorder.

Genetic tests is another diagnostic tool that suggested to general population and in individual cases adapted to genetic diseases that are known.

In 2008 about 75.5% of the population in Israel were Jews, 20.2% Arabs, and 4.3 were defined as "others". Approximately 45% of Arabs living in the northern region compared to 10% of the Jewish population. Congenital malformations were the leading cause of death in infants Arab and the second cause of death in Jewish infants.

In recent years the supply of screening before and during pregnancy has increased, but it is apparent that the rate of implementation of nuchal translucency, amniocentesis and therefore detection of disease are lower in Arab population, as well as the rates of taking folic acid. These differences between populations in carrying out tests that enable prevention and early detection of birth defects and neonatal genetic diseases also associated with differences in economic, religious and age of the woman.

In this work we try to know the population applying for medical services at Hillel Yaffe Hospital. Estimate the rate of risk factors for appearance of disease or fetal malformations in a population who turn to hospital "Hillel Yaffe" and examine whether there is a difference in the rate of early testing for diseases or birth defects in the fetus.

We hypothesize that a large percentage of the population who turn to Hillel Yaffe Hospital has risk factors for having a sick fetus and the Muslim population is in higher risk than the Jewish population.

Understanding the population and its risk factors, will allow specific reference to these risk factors to lowering them to eventually reduce the rate of congenital malformations in this population.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who address the emergency room, Ultrasound unit or foreign clinics in the second or third trimester.

Exclusion Criteria:

* Pregnant women in the first trimester Pregnant women who doesn't want to participate.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women who address the emergency room, Ultrasound unit or foreign clinics.
Sampling Method: Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2012-08; Primary Completion 2012-09 (Estimated); Study Completion 2013-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: yael yagur, student, Principal Investigator — Technion, Israel Institute of Technology; Alon Shrin, M.D., Study Director — Ultrasound unit manager, obstetric and gynaecology, Hillel Yaffe
Locations (1):
- Obstetric and Gynaecology Department, Hadera, Israel